CLINICAL TRIAL: NCT01281358
Title: Development and Evaluation of a Parenting Intervention to Promote Development in Infants Born Very Premature
Brief Title: Helping Our Premature Infants ON to Better Motor Skills (HOP-ON)
Acronym: HOP-ON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Action Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 10027
Record Dates: First submitted 2011-01-05; First posted 2011-01-21 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Motor Development of Premature Infants
Keywords: Premature infants; Motor Development
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOP-ON intervention (Experimental): Participants will receive a CD-ROM (or DVD and booklet if no access to computer) highlighting motor skills which could be encouraged with premature infants
  Interventions: Other: HOP-ON
- SMILES (Active Comparator): Participants will received a CD-ROM (or DVD and booklet if no access to a computer) which contains information on interacting with their premature infant
  Interventions: Other: SMILES

INTERVENTIONS:
Other: HOP-ON — A programme of activities which promote motor development
  Arms: HOP-ON intervention
Other: SMILES — Details are provided on ways for parents to interact with their premature infants
  Arms: SMILES

SUMMARY:
Infants born very premature have biological risk factors for later developmental coordination disorder. Parental stereotyping of infants as fragile and other environmental factors, such as spending long periods laying on their backs, also contribute to motor delay. This study aims to develop and evaluate a computer-based intervention (Helping Our Premature infants ON to better motor skills - HOP-ON) for parents of preterm infants. HOP-ON will model evidence based strategies to develop infants' fine and gross motor skills, and aims to reduce parental stereotyping. It is hypothesised that infants whose parents receive the HOPON CD-ROM/DVD and Booklet will have better motor skills at 12 months adjusted age compared to those whose parents receive a control CD-ROM/DVD and booklet. Parents of infants born at less than 32 weeks gestation (target n = 138) will be recruited prior to discharge from the neonatal unit and randomised to either HOP-ON or control. The primary outcome is motor score (Bayleys III) at 12 months adjusted age. Other outcomes are parental confidence and perceptions of infant capability at 3 months and quality of movement, infant growth, fine and gross motor movement and parenting stress at 12 months. Data will be analysed blind to study condition and on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born less than 32 weeks of gestation, and progressing well enough to have either been recently discharged from hospital, or being discharged from hospital within the next two weeks.
* Parent/s aged between 16-60 years of age, who have a preterm infant - born less than 32 weeks of gestation.

Both parent and infant inclusion criteria must be met for inclusion in the study.

Exclusion Criteria:

* Parent/s of infants who are still receiving hospital care at 3 months adjusted age, and their premature infants who are still receiving hospital care at 3 months adjusted age.
* Parent/s of multiple births, where the number of infants is greater than two (three of more infants).
* To avoid excessive travel costs, infants born outside the defined catchment area will be excluded from the study. There are no other exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Difference in Bayley III motor scales scores | 12 months corrected age

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Derby Hospitals NHS Foundation Trust, Derby
  - University Hospitals Leicester NHS Trust, Leicester
  - Nottingham University Hospitals NHS Trust, Nottingham